CLINICAL TRIAL: NCT04787016
Title: Effects of Pilates Training on Physical Performance of Cricketers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Principal Investigator, Waqar Ahmed Awan, Professor, Riphah International University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Ramsha
Record Dates: First submitted 2021-02-20; First posted 2021-03-08 (Actual); Last update posted 2021-03-08 (Actual); Status verified 2021-03

CONDITIONS: Core Strengthening

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pilate training (Experimental): The participants of this group perform pilate training along with conventional cricket training.
  Interventions: Other: Pilate training
- Conventional training (No Intervention): The participants perform only conventional cricket training.

INTERVENTIONS:
Other: Pilate training — Pilates is an exercise training program used to build core strength and flexibility.
  Arms: Pilate training

SUMMARY:
This study is designed to evaluate the effectiveness of Pilates training improves physical fitness of cricket players.

DETAILED DESCRIPTION:
During the modern times, researchers have notably increased their knowledge, grounded on literature, with regards to the relationship between core stability and athletic performance. Number of research studies have also been completed that underline the benefits of core stability training on injury prevention or performance, but in combination with other training modalities such as speed, power, strength and agility. Although several studies have investigated core stability benefits in athletes but there are very limited studies have presented the role of Pilate training in increasing the core strength and stability of cricket players in order to maximize their performance in the game. This study will contribute in describing the effects of Pilate training in cricket players.

ELIGIBILITY:
Inclusion Criteria:

* Participants falling in this category would be recruited into the study. Active Male cricketers. Had practiced for at least 2 years Age group of 19-30 Players with normal BMI (ranging in between 18.5 to 24.9)

Exclusion Criteria:

* Participant failing to fall in this category would be excluded of the study. History of metabolic diseases.

History of recent fractures. Players taking substance inhibited (in and out of the competition) by WADA Had extreme discomfort on contracting the abdominal muscles.

Were spin bowlers.

Ages: 19 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Self representation
Enrollment: 20 (Estimated)
Dates: Start 2020-06-10 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-03-30 (Estimated)

PRIMARY OUTCOMES:
To evaluate the effectiveness of Pilates training improves physical fitness of cricket players. | 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Riphah international University, Islamabad, Federal, Pakistan